CLINICAL TRIAL: NCT06027775
Title: Chemotherapy Alone Versus Chemotherapy Plus Targeted Therapy as Adjuvant Therapy for Initially Unresectable Colorectal Cancer Liver Metastases: A Retrospective Cohort Study
Brief Title: Chemotherapy Alone Versus Chemotherapy Plus Targeted Therapy as Adjuvant Therapy for Initially Unresectable Colorectal Cancer Liver Metastases
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Head of Colorectal Surgery, Fudan University
Other Study IDs: CAPTIUM
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chemotherapy plus Targeted therapy (CT): The treatment decisions and evaluation of treatment outcomes, such as the assessment of metastases resectability and tumor response, were carried out by the multi-disciplinary team (MDT) comprising experts from each medical centers. In this cohort, initially unresectable colorectal cancer liver metastasis (CRLM) patients who were successfully converted and achieved no evidence of disease status were treated with chemotherapy plus targeted therapy, as adjuvant therapy.
  Interventions: Drug: Targeted agent
- Chemotherapy Alone (CA): In this cohort, initially unresectable colorectal cancer liver metastasis (CRLM) patients who were successfully converted and achieved no evidence of disease status were treated with chemotherapy, as adjuvant therapy.

INTERVENTIONS:
Drug: Targeted agent — The two cohorts received different adjuvant therapy regimens, with the CT group receiving chemotherapy plus targeted therapy; the CA group received chemotherapy alone.
  Groups: Chemotherapy plus Targeted therapy (CT)

SUMMARY:
Chemotharapy plus targeted therapy regimen, as an adjuvant therapy, can effectively reduce the rate of both intrahepatic and extrahepatic recurrence in initially unresectable CRLM patients. Those with KRAS/NRAS/BRAF mutated tumors or cycle of conversion therapy ≤ 4 can benefit more from chemotharapy plus targeted therapyrather than from chemotharapy alone, with a tolerable toxicity profile.

DETAILED DESCRIPTION:
This multi-center study enrolled consecutive patients with initially unresectable CRLM who underwent conversion therapy or radiofrequency ablation (RFA) and achieved no NED status between June 1, 2013, and June 30, 2020, from Zhongshan Hospital of Shanghai, Zhongshan Hospital of Xiamen, Cancer Hospital of Beijing. The inclusion criteria were as follows: (1) with histologically confirmed CRC; (2) with initially unresectable synchronous liver metastases (LMs); (3) accepted conversion therapy and successfully converted into resectable status; (4) underwent R0 intestinal and hepatic resection; (5) accepted adjuvant therapy. The exclusion criteria were as follows: (1) R1/R2 resection; (2) extrahepatic metastases; (3) accepted postoperative monotherapy; (4) lack of follow-up data. According to the adjuvant therapy regimen (with or without targeted therapy), the cohorts were divided into CA cohort and CT cohort. The study was approved by the ethics committee of three medical centers and was adhered to Good Clinical Practice guidelines and the Declaration of Helsinki. Written informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years;
2. Histologically confirmed CRC;
3. Initially unresectable synchronous liver metastases (LMs);
4. Accepted conversion therapy and successfully converted into resectable status;
5. Underwent R0 intestinal and hepatic resection;
6. Accepted adjuvant therapy.

Exclusion Criteria:

1. R1/R2 resection;
2. Extrahepatic metastases;
3. Accepted postoperative monotherapy;
4. Lack of follow-up data.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Initially unresectable CRLM patients who were successfully converted and achieved no evidence of disease status from June 2013 to June 2020 were retrospectively collected. 1:2 propensity score matching (PSM) was performed to balance the baseline characteristics between CA and CT cohorts. After PSM, 196 patients werethe disease-free survival (DFS) and overall survival (OS) were evaluated between two cohorts （CA:N=66, CT:N=132）.
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
relapse-free survival | 3 years
  The relapse-free survival (PFS) was defined as the period from the start of initial liver resection to the date of tumor relapse or death

SECONDARY OUTCOMES:
overall survival | 5 years
  The overall survival (OS) was defined as the period from the start of initial liver resection until death from any cause, at which point the data was censored.

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, MD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No